CLINICAL TRIAL: NCT05961358
Title: Auxiliary Anesthesia Technique for Extracting Advanced Hemodynamic Parameters Based on Peripheral Arterial Waveform Photography
Status: Active, not recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0554
Record Dates: First submitted 2023-07-06; First posted 2023-07-27 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia
Keywords: arterial blood pressure; cardiac output; advanced hemodynamic; mobile Applications
MeSH Terms: interventions — Transducers, Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General anesthesia Patients: Subjects experiencing general anesthesia
  Interventions: Procedure: snapshots or videos of monitor; Procedure: Pressure transducer

INTERVENTIONS:
Procedure: snapshots or videos of monitor — The mobile device（a phone）was used to obtain the screen image of the monitor, and the arterial blood pressure waveform is extracted by image processing technology.
Procedure: Pressure transducer — Arterial catheter were connected to conventional pressure transducers and Flotrac-Vigileo transducers.

SUMMARY:
In this study, the arterial blood pressure waveform was digitized by snapshots or videos of the patient monitor to further estimate advanced hemodynamic parameters, so as to realize continuous and automatic monitoring of advanced hemodynamics on mobile devices to assist anesthesia, with a view to developing an Android/iOS application for mobile devices and application in patient management.

ELIGIBILITY:
Inclusion Criteria:

* Invasive blood pressure monitoring
* Aged 18-65 years
* ASA class I-III

Exclusion Criteria:

* Spontaneous breathing
* Prone position
* Non-radial artery cannulation
* Aortic regurgitation
* Heart arrhythmia
* Heart rate > 100/min
* Intra-aortic balloon pump
* Peripheral vascular disease
* Body weight < 40 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at the Second Affiliated Hospital Zhejiang University School of Medicine. The study participants will be adult general anesthesia patients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of mobile device analysis results with Vigileo analysis results | 1 day
  Cardiac output and Stroke Volume Variation were acquired by mobile device and Vigileo
Comparison of arterial waveform collected directly analysis results and Vigileo analysis results | 1 day
  Cardiac output and Stroke Volume Variation were acquired by Vigileo and arterial waveform collected directly analysis
Comparison of arterial waveform collected directly analysis results and mobile device analysis results | 1 day
  Cardiac output and Stroke Volume Variation were acquired by mobile device and arterial waveform collected directly analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No